CLINICAL TRIAL: NCT04237961
Title: Ancillary Procedures in Patients of Refractory Facial Palsy Patients Selection and Evaluation of the Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, saleh ali ibrahim elazoumi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Assiutu123
Record Dates: First submitted 2018-03-25; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Facial Palsy
MeSH Terms: conditions — Facial Paralysis | interventions — Botulinum Toxins, Type A; Injections; Sutures

STUDY DESIGN:
Intervention Model Description: Patients could be divided into three groups according to the anatomical site of interferences:
  * Group 1: Upper third interferences
  * Group 2: Mid third interferences
  * Group 3: Lower third interferences
Who Masked: Participant
Masking Description: Patients could be divided into three groups according to the anatomical site of interferences:
  * Group 1: Upper third interferences
  * Group 2: Mid third interferences
  * Group 3: Lower third interferences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper third interference (Experimental): Botox & brow lift
  Interventions: Procedure: Botox and brow lift
- Middle third (Experimental): Botox and fat injection
  Interventions: Procedure: Injection
- Lower third (Experimental): Suspension suture
  Interventions: Procedure: Suture

INTERVENTIONS:
Procedure: Botox and brow lift — Botox injection
  Arms: Upper third interference
Procedure: Injection — Fat injection and botox
  Arms: Middle third
Procedure: Suture — Suspension suture
  Arms: Lower third

SUMMARY:
Introduction:

There are numerous causes of facial palsy (FP), though hemifacial weakness is often generally termed Bell's palsy, named after the Scottish neurologist Charles Bell, who described sudden onset unilateral facial paralysis in 1821.

Virally triggered, acute FP, to which the term Bell's palsy (BP) refers, is one of the most common, and fortunately the most likely condition to result in eventual return to premorbid status; 70% to 90% of patients recover spontaneously. Other causes of FP routinely result in poorer recovery, and the clinician must discern among these to formulate a treatment plan.

In facial palsy, paralysis of muscles on the affected side of the face results in loss of forehead creases, loss of the nasolabial fold, lagophthalmos, brow droop, and drooping of the corner of the mouth. In contrast, muscles on the unaffected side of the face no longer have opposing forces.

This may cause difficulty in articulation, eating, drinking, and is often cosmetically unacceptable to patients because of asymmetry, especially when speaking, smiling, and laughing. There are significant psychological effects as patients lack the confidence to carry out many daily activities in public, such as appearing in photographs.

Although management is difficult, there are a range of reanimation options available. These include nerve grafts, muscle transfers, myofunctional approaches, and microsurgical patches usually for the more severe facial palsies (House-Brackmann grades 4 to 6). However, despite these procedures, facial symmetry may not improve.

DETAILED DESCRIPTION:
Ancillary procedures in patients of refractory facial palsy. Patients selection and evaluation of the outcomes.

Introduction:

There are numerous causes of facial palsy (FP), though hemifacial weakness is often generally termed Bell's palsy, named after the Scottish neurologist Charles Bell, who described sudden onset unilateral facial paralysis in 1821.

Virally triggered, acute FP, to which the term Bell's palsy (BP) refers, is one of the most common, and fortunately the most likely condition to result in eventual return to premorbid status; 70% to 90% of patients recover spontaneously. Other causes of FP routinely result in poorer recovery, and the clinician must discern among these to formulate a treatment plan.

In facial palsy, paralysis of muscles on the affected side of the face results in loss of forehead creases, loss of the nasolabial fold, lagophthalmos, brow droop, and drooping of the corner of the mouth. In contrast, muscles on the unaffected side of the face no longer have opposing forces.

This may cause difficulty in articulation, eating, drinking, and is often cosmetically unacceptable to patients because of asymmetry, especially when speaking, smiling, and laughing. There are significant psychological effects as patients lack the confidence to carry out many daily activities in public, such as appearing in photographs.

Although management is difficult, there are a range of reanimation options available. These include nerve grafts, muscle transfers, myofunctional approaches, and microsurgical patches usually for the more severe facial palsies (House-Brackmann grades 4 to 6). However, despite these procedures, facial symmetry may not improve.

Refractory Facial Palsy:

Facial paralysis is a rare disorder, but it has significant effects on an individual, both physical and emotional. While most patients fully recover from acute facial paralysis, a small population is left with chronic lingering symptoms. Refractory patients are those who had the maximum benefit of a performed procedure and need some fine touches and also those who did not recover well of the initial condition.

Aim of the Work:

This study is aimed to evaluate the outcome of ancillary procedures in refractory cases of facial palsy and to introduce both simple and sophisticated techniques to those patients presented to the investigator's department.

Inclusion Criteria:

Patients with refractory Facial Palsy who did not respond well to other concerned interferences and those who presented the maximum benefit possible of a performed procedure.

Patients & Methods:

This study will be conducted on 20 patients attendance outpatient clinic of plastic surgery department - Assiut University Hospital.

Patients could be divided into three groups according to the anatomical site of interferences:

* Group 1: Upper third interferences
* Group 2: Mid third interferences
* Group 3: Lower third interferences Methodology
* Botulinum toxin A (BTXA) has been used since the 1970s to treat a variety of conditions resulting in abnormal muscle contraction or spasm. It works by preventing the release of acetylcholine into the neuromuscular junction thereby inhibiting muscle contraction.2 Its benefits in synkinesis in facial palsy (aberrant neural regeneration of the paralysed muscles) are well recognized.

BTXA was injected into the contralateral lower facial muscles complex to weaken the unopposed normal muscles to improve symmetry, both active and passive.

• Gold/Platinum weight implants Implantable devices have been used to restore dynamic lid closure in cases of severe, symptomatic lagophthalmos. These procedures are best for patients with poor Bell phenomenon and decreased corneal sensation. Gold or platinum weights, a weight-adjustable magnet, or palpebral springs can be inserted into the eyelids. Pretarsal gold-weight implantation is most commonly performed.

The implants are inert and composed of 99.99% pure gold or platinum. Sizes range from 0.6-1.8 g. The weight allows the upper eyelid to close with gravity when the levator palpebrae are relaxed. Therefore, patients must sleep with their head slightly elevated.

The implants are easily removed if nerve function returns. Complications include migration of the implant, inflammation, allergic reaction, and extrusion.

• Tarsorrhaphy Tarsorrhaphy decreases horizontal lid opening by fusing the eyelid margins together, increasing support of the precorneal lack of tears and improving coverage of the eye during sleep. The procedure can be done in the office and is particularly suitable for patients who are unable or unwilling to undergo other surgery.

Tarsorrhaphy can be performed laterally, centrally, or medially. The lateral procedure is the most common; however, it can restrict the monocular temporal visual field.

* Brow lifting Brow ptosis is repaired with a direct brow lift. Care should be taken in the presence of corneal decompensation because lifting the brow can cause worsening of lagophthalmos, especially if lid closure is poor. A gold-weight implant can be placed or lower-lid resuspension can be performed simultaneously to prevent this complication
* Suspension suture Static facial suspension procedures stabilise the muscles of mid-face paralysis and provide facial symmetry, a better aesthetic appearance, improved chewing and speech production in patients with facial paralysis. The new generation of Silhouette wires for tissue suspension is a significant improvement with respect to gold threads or Russian threads. They provide a new method of anchoring since they are made of polypropylene with absorbable cones of polylactic acid and glycolic acid. This suture allows tissue growth in and around the cones and therefore a strangerhood.

They were approved by the FDA in November 2006 and by the EEC in March 2007. They have been used in over 6,000 mid-face facial aesthetic surgery interventions in the U.S. and Europe and have recently begun to be used to treat facial paralysis.

* Fat injection Fat transfer to the face uses the patient's own adipose tissue (collected with a minor liposuction procedure from the belly or back), which gives volume and shape to the affected parts of the face, as well as impart glow and sheen to the skin
* Lateral Canthoplasty:

canthoplasty may be considered as one of the most valuable oculoplastic surgical procedures to correct lid abnormalities. The indications include ectropion, entropion, lateral canthal dystopia, horizontal lid laxity, lid margin eversion.

Evaluation of outcome:

-Subjective:- 3 Plastic surgeon will be commenting on the pre and post photography regarding to normal side .

-Objective:- measurement between normal and effected side of the position eye brow ,Palpebral fissure, and angle of the mouth

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory Facial Palsy who did not respond well to other concerned interferences and those who presented the maximum benefit possible of a performed procedure.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-28 (Estimated); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Ancillary Procedures in Patients of Refractory Facial Palsy Patients Selection and Evaluation of the Outcomes | 2 years
  measurement the change in vertical length of the palpebral fissure of the affected eye before and after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No
Patients Selection and evaluation of the outcome.